CLINICAL TRIAL: NCT06341803
Title: Personalized Transcranial Magnetic Stimulation Treatment for Depression
Acronym: APIC-TMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mental Health, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB 2023/00397
Record Dates: First submitted 2024-01-22; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Depression
Keywords: neuronavigated; iTBS; Accelerated
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Individually neuronavigated intermittent theta burst stimulation (Magpro X100) system for depression (Experimental): Participants will receive an accelerated intermittent theta burst stimulation (iTBS) treatment delivered with a MagVenture MagPro X100 system (MagVenture A/S, Denmark) equipped with a butterfly shaped MagVenture Cool-B65 A/P coil. The treatment course is comprised of 10 treatment sessions daily for 5 consecutive workdays for a total of 50 sessions. Each iTBS session is approximately 10 minutes (depth corrected Resting Motor Threshold of 90%, 60 cycles of 10 bursts of three pulses at 50 Hz, repeated at 5 Hz; 2s on and 8s off; 1800 pulses per session; with a 50-minute interval between sessions). All iTBS sessions will be performed by staff trained and credentialed in TMS according to Singapore College of Psychiatrists guidelines.
  Interventions: Device: Individually Neuronavigated accelerated intermittent theta burst stimulation with Magpro X100

INTERVENTIONS:
Device: Individually Neuronavigated accelerated intermittent theta burst stimulation with Magpro X100 — MagproX 100 and Axilium Cobot with Localite camera

SUMMARY:
This proposal seeks to conduct a pragmatic single arm, open label pilot implementation to validate our individualized functional Magnetic Resonance Imaging (fMRI) connectome-guided localization approach for accelerated TMS among Asian patients with depression.

Participants will be patients with Major Depressive Disorder not responding to standard treatment, with no exclusions to fMRI or transcranial magnetic stimulation (TMS) (essentially metal implants in the head) and willing to participate in the pilot.

All participants will undergo MRI scans before and after the accelerated TMS treatment. The multi-session hierarchical Bayesian model (MS-HBM) approach will be used to estimate individualized connectome-guided target locations.

Patients will undergo accelerated TMS applied to individualized connectome-guided target locations (based on the MS-HBM approach).

Patients will undergo 10 sessions (each session lasting 10 min) spread out over 10 hours each day for 5 consecutive working days.

All clinical outcome data will be collected for each patient by a pre-defined questionnaire at four time points: at baseline, post-treatment, 1 month and 3 months during follow-up.

The clinical outcome data will be analyzed using linear regression or repeated analysis of variance (ANOVA) after adjusting for baseline clinical characteristics and socio-demographics. Trajectories of the clinical outcome data at baseline, post-treatment and all follow-up time points will be plotted and compared with time series statistical analysis models with the other clinical and socio-demographic characteristics included as confounders.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years.
2. DSM-5 diagnosis of current Major Depressive Episode.
3. Montgomery-Asberg Depression Rating Scale score of 20 or more.
4. Inadequate response to an adequate trial (4 weeks) of at least one antidepressant medication.
5. Able to give informed consent.

Exclusion Criteria:

1. DSM-5 psychotic disorder
2. Drug or alcohol abuse or dependence (preceding 3 months).
3. Rapid clinical response required, e.g., high suicide risk.
4. Significant neurological disorder, which may pose increased risks with TMS, e.g., epilepsy.
5. Metal in the cranium, skull defects, pacemaker, cochlear implant, medication pump or other electronic device.
6. Pregnancy.
7. Unsuitable for MRI.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline, immediately post treatment, 1 month and 3 months post intervention
  Clinician rated Depression rating scale, range of scores 0 to 60 with higher scores meaning a worse outcome

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology (16-Item) (Self-Report) (QIDS-16) | Baseline, (Days 1-5 of treatment), immediately after intervention, 1 month and 3 months post intervention
  Patient rated Depression rating scale, scored 0-27 with higher scores meaning a worse outcome
Montreal Cognitive Assessment (MoCA), | Baseline, immediately post treatment, 1 month and 3 months post intervention
  global cognitive functioning, scored 0 to 30 with higher scores meaning better outcome
EuroQol- 5 Dimension (EQ-5D) | Baseline, immediately post treatment, 1 month and 3 months post intervention
  Quality of life scales, Visual analogue scale 0-100 with higher scores meaning better outcome
Quality of Life Enjoyment and Satisfaction Questionnaire Short form (Q-LES-QS-SF) | Baseline, immediately post treatment, 1 month and 3 months post intervention
  Quality of life scales, scored 0-70 with higher scores meaning better outcome

OTHER OUTCOMES:
Correlation of changes in functional connectivity with changes in MADRS scores | Baseline, immediately post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Mental Health, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No